CLINICAL TRIAL: NCT05273112
Title: Evaluation of the Variation in Quality of Life During Medical Transition According Different Modalities of Supported Care for Transgender People.
Brief Title: Evaluation of the Variation in Quality of Life During Medical Transition for Transgender People.
Acronym: TRANS'ITION
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_09; 2021-A00154-37 (Other: ID-RCB number, ANSM); PREPS-19-0078 (Other: AAP number, DGOS)
Record Dates: First submitted 2021-12-24; First posted 2022-03-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-11

CONDITIONS: Gender Dysphoria
Keywords: Transidentity; Gender Dysphoria; Transition; Quality of Life
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transgender people can benefit from psychological, psychiatric, endocrinological support, sexual reassignment surgery, sexology support and dermatological care. The value of transitional care courses is scientifically recognized. Currently, the modalities of decision and realization of the care paths are heterogeneous on the territory, little standardized, and are the subject of debates between representatives of users and medical teams.

The french national report of IGAS from 2011 warns of the need to argue and legitimize care practices through more numerous, more exhaustive scientific studies, presenting a better level of evidence

Since 2011, no prospective study has been carried out on the national and international level, making it possible to assess the relevance of the planned care modalities. This research project, conducted over five consecutive years at the first contact of a transgender people with a care device, aims to correlate a variation in the quality of life of people with the characteristics of the care methods provided. This is a first proposal to assess care practices for transgender people. The results of this study would first allow us to infer the care modalities most suited to the needs of people. Secondly, secondary hypotheses could support new experimental protocols.

DETAILED DESCRIPTION:
This research is a prospective multicenter cohort study with a 3-year and 5-year follow-up of transgender people in medical transition.

Main aim:

Evaluate the evolution of the quality of life during five years in transgender people who benefit from transition support cares.

Secondary objectives:

Secondary objective n°1 :

Identify the different factors that influence the evolution of quality of life evaluated over three years in transgender people who benefit from transition support cares.

Secondary objective n°2 :

Evaluate the evolution of the satisfaction of the shared medical decision for transgender people in medical transition.

Secondary objective n°3 :

Evaluate the evolution of the satisfaction of body image for transgender people in medical transition.

Secondary objective n°4 :

Evaluate the evolution of psychiatric comorbidities for transgender people in medical transition.

Secondary objective n°5 :

Evaluate the benefits and limits in long term (five years) on the quality of life, the satisfaction of the shared medical decision, the satisfaction of body image and the evolution of psychiatric comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of Gender Dysphoria according to DSM5 diagnostic criteria
* Wishing to benefit from supportive care for their transition trajectory and addressing a care system represented by the collaborating centers participating in the study,
* Willing to comply with all study procedures and duration,
* Understanding and able to speak French.

Exclusion Criteria:

* Minor or adult under curatorship, under judicial protection, persons deprived of their liberty
* Refusal to participate after clear and fair information from the study
* Person with sexual reassignment surgery or with cross hormon therapy since two years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: transgender people in medical transition
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores | 3 years
  Scores on the WHOQOL BREF (World Health Organisation Quality Of Life) scale

SECONDARY OUTCOMES:
Social factors (age, gender, profession, knowledge of care system) | Baseline and 6 months, 12 months, 18 months, 24 months, 30 months, 3 years and 5 years
  Answers given by the patient during interview
Satisfaction of the shared medical decision | 6 months, 12 months, 18 months, 24 months, 30 months, 3 years and 5 years
  Scores on the CDIS (Clinical Decision-making Involvement and Satisfaction) clinical decision making involvement and satisfaction score 15 questions scored 1-5 (totally disagree, strongly disagree, neither agree nor disagree, strongly agree, totally agree)
Satisfaction of body image | 6 months, 12 months, 18 months, 24 months, 30 months, 3 years and 5 years
  Score on the BIS (Body Image Scale), total score ranges from 0 to 30, A higher score means a higher level of body image disturbance
General psychopathology | 6 months, 12 months, 18 months, 24 months, 30 months, 3 years and 5 years
  French version of Mini International Neuropsychiatric Interview (DSM)
Anxiety and depression | 6 months, 12 months, 18 months, 24 months, 30 months, 3 years and 5 years
  Anxiety and depression scores on the HAD scale (Hospital Anxiety and Depression scale), a score upper 8 means is considered as a risk of an anxiety or depressive disorder
Quality of life scores | 6 months, 12 months, 18 months, 24 months, 30 months, 5 years
  Scores on the WHOQOL BREF (World Health Organisation Quality Of Life) scale

CONTACTS AND LOCATIONS:
Overall Officials: François MEDJKANE, MD, Principal Investigator — University Hospital, Lille
Locations (13):
- France (13):
  - Centre Hospitalier de Béziers, Béziers
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CHU de Lille, Lille
  - Maison de Santé Lille Moulins, Lille
  - Maison de Santé Lille Sud, Lille
  - CHU de Lyon, Lyon
  - G..R.E.T.T.I.S, Lyon
  - Hopital de la Conception - Marseille, Marseille
  - CHU de Nice, Nice
  - Centre Hospitalier Maison Blanche, Paris
  - Centre Hospitalier Sainte-Anne, Paris